CLINICAL TRIAL: NCT06940102
Title: A Multicenter, Real-World Study on Nano-Crystalline Megestrol Acetate for Cachexia in Patients With Advanced Digestive System Tumors Receiving TKI-Based Therapy
Brief Title: Real-World Study on Nano-Crystalline Megestrol Acetate for Cachexia in TKI-Treated Advanced Digestive Tumors
Status: Recruiting | Type: Observational
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MGA-DSC-601
Record Dates: First submitted 2025-03-26; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Cachexia; Digestive System Cancer; Gastric Cancer; Colorectal Cancer; Hepatocellular Carcinoma
Keywords: Megestrol Acetate; Nano-crystalline Megestrol Acetate; Targeted Therapy; Tyrosine Kinase Inhibitors; Prospective Studies; Observational Studies; Antineoplastic Agents; Digestive System Cancer
MeSH Terms: conditions — Cachexia; Digestive System Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nano-crystalline Megestrol Acetate Oral Suspension +TKI-Based Therapy: Nano-crystalline Megestrol Acetate Oral Suspension, with a specification of 125 mg/mL, the study group takes 5 mL orally per day (625 mg/day)，TKI Therapy ± chemotherapy / immunotherapy
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Drug: TKI-Based Therapy
- TKI-Based Therapy: TKI Therapy ± chemotherapy / immunotherapy
  Interventions: Drug: TKI-Based Therapy

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nano-crystalline Megestrol Acetate Oral Suspension, with a specification of 125 mg/mL, the study group takes 5 mL orally per day (625 mg/day)
  Groups: Nano-crystalline Megestrol Acetate Oral Suspension +TKI-Based Therapy
Drug: TKI-Based Therapy — TKI-Based Therapy

SUMMARY:
This study is a prospective, observational clinical study aimed at evaluating the efficacy of Megestrol Acetate for cachexia in patients with advanced digestive system tumors receiving TKI-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign a written informed consent (ICF).
* Age ≥ 18 years at enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy ≥ 3 months.
* Histologically or cytologically confirmed locally advanced or metastatic digestive system tumors that are not amenable to curative treatment, according to the 8th edition TNM staging classification.
* Not benefiting from local anticancer therapies such as surgery, local ablation, or chemoembolization, and planned to receive TKI-based anticancer treatment, which may be combined with chemotherapy or immunotherapy).
* Meet the diagnostic criteria for pre-cachexia or cachexia (based on Fearon diagnostic criteria).
* Good organ function determined

Exclusion Criteria:

* Gastrointestinal obstruction.
* Anorexia due to difficulty in eating caused by neurosis, mental illness, or pain.
* Comorbidities such as severe cerebrovascular, cardiac, renal, or liver diseases.
* Major surgery or trauma within the last month.
* Allergy to any component of the investigational drug.
* Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic digestive system tumors
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Appetite improvement level | From baseline to Week 12 (end of treatment period)
  Proportion of subjects with an improvement in appetite based on A/CS-12 after 12 weeks of treatment
Weight improvement level | From baseline to Week 12 (end of treatment period)
  Proportion of subjects who did not lose weight relative to baseline after 12 weeks of treatment

SECONDARY OUTCOMES:
progression-free survival (PFS) | From the date of randomization until the first documented disease progression or death from any cause, whichever occurs first，assessed up to 24 months
  defined as the duration from the start treatment to progression, or patient death

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Du, Principal Investigator — The General Hospital of Northern Theater Command; Zhenguang Du, Principal Investigator — Organizational Affiliation: Liaoning Cancer Hospital
Locations (2):
- China (2):
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning